CLINICAL TRIAL: NCT00035386
Title: Trans-Right Ventricular Approach to Alcohol Septal Ablation in Obstructive Hypertrophic Cardiomyopathy: A Pilot Feasibility Study
Brief Title: Alcohol Septal Ablation in Obstructive Hypertrophic Cardiomyopathy: A Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020125; 02-H-0125
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-04

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Outflow Obstruction; ICE; HCM; Hypertrophic Cardiomyopathy; OHC; Obstructive HCM; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathies | interventions — Ethanol

INTERVENTIONS:
Procedure: trans-right ventricular alcohol septal ablation (TRVASA)

SUMMARY:
This study will test the feasibility of a modified procedure for treating obstructive hypertrophic cardiomyopathy (OHC). Patients with OHC have a thickening of the heart muscle that obstructs blood flow out of the heart, causing breathlessness, chest pain, palpitations, tiredness, lightheadedness, and fainting.

The current treatment for OHC is a procedure called alcohol septal ablation (also percutaneous transluminal septal ablation, or PTSA), which involves injecting a small amount of alcohol into a tiny artery that supplies the part of muscle causing blood flow obstruction. The success of PTSA is limited, however, by problems of heart anatomy and the ability to find the appropriate artery to inject. Modifying the procedure by injecting the alcohol through the wall of the lower right chamber of the heart may improve its safety and effectiveness. The new technique requires positioning a catheter (a flexible tube) into the appropriate area of the heart. This study will test the ability to accurately guide the catheter to that area.

Patients with OHC 18 years of age and older who are scheduled to have a cardiac catheterization may be eligible for this study. At the end of the catheterization procedure, participants will undergo intra-cardiac echocardiographic imaging. For this test, one of the catheters placed in the femoral artery (at the top of the leg) for cardiac catheterization will be substituted for a larger one. Through this catheter, a special catheter will be introduced and advanced to the heart to provide images. This pilot feasibility study does not involve injection of alcohol.

DETAILED DESCRIPTION:
Patients with obstructive hypertrophic cardiomyopathy (HCM) and drug-refractory symptoms have traditionally been referred for cardiac surgery to widen the left ventricular (LV) outflow tract. More recently, percutaneous transluminal septal ablation (PTSA) has also been shown to thin the subvalvular septum and thereby to reduce LV outflow pressure gradients and to improve symptoms in obstructive HCM. However, this procedure is not infrequently limited by septal coronary artery anatomy and inability to identify and cannulate the appropriate artery that supplies the septal region of interest. Some attempts are also associated with coronary artery dissection, particularly, if there is associated coronary artery disease. A trans-right ventricular (RV) alcohol septal ablation (TRVASA) would significantly simplify the procedure, and increase its safety. The purpose of this study is to initially test our ability to visualize and guide a delivery catheter to a targeted part of the anterior interventricular septum involved in the generation of the LV outflow obstruction using intracardiac echocardiography (ICE). No therapy is intended: alcohol will not be injected into the septum in this initial study.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients of either gender, aged 18-85 years.

Symptomatic patients receiving clinically indicated evaluation for cardiomyopathy and found to have obstructive HCM.

LV outflow tract gradient greater than 30 mm Hg at rest by echocardiography or cardiac catheterization.

EXCLUSION CRITERIA:

Positive pregnancy test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12
Dates: Start 2002-04; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] McIntosh CL, Maron BJ. Current operative treatment of obstructive hypertrophic cardiomyopathy. Circulation. 1988 Sep;78(3):487-95. doi: 10.1161/01.cir.78.3.487. No abstract available. PMID 3409494
- [Background] Krajcer Z, Leachman RD, Cooley DA, Coronado R. Septal myotomy-myomectomy versus mitral valve replacement in hypertrophic cardiomyopathy. Ten-year follow-up in 185 patients. Circulation. 1989 Sep;80(3 Pt 1):I57-64. PMID 2766539
- [Background] Delahaye F, Jegaden O, de Gevigney G, Genoud JL, Perinetti M, Montagna P, Delaye J, Mikaeloff P. Postoperative and long-term prognosis of myotomy-myomectomy for obstructive hypertrophic cardiomyopathy: influence of associated mitral valve replacement. Eur Heart J. 1993 Sep;14(9):1229-37. doi: 10.1093/eurheartj/14.9.1229. PMID 8223738